CLINICAL TRIAL: NCT00134992
Title: Single-Center, Randomized, Double Masked, Two-Period Cross-Over, Three Days Per Period, Phase IV Study to Compare Ocular Safety and Tolerability of Prednisolone Acetate 0.5% Eye Drops Versus Vehicle in Healthy Volunteers
Brief Title: A Study to Compare Ocular Safety and Tolerability of Prednisolone Acetate 0.5% Eye Drops Versus Vehicle in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CULT 491 DE 02
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2006-06-09 (Estimated); Status verified 2006-06

CONDITIONS: Healthy
Keywords: Prednisolone acetate; eye drops; tolerability; Healthy volunteers
MeSH Terms: interventions — prednisolone acetate

INTERVENTIONS:
Drug: Prednisolone acetate

SUMMARY:
The objective of this trial was to confirm the tolerability of prednisolone acetate 0.5% eye drops by testing the hypothesis that the ocular safety and tolerability of prednisolone acetate 0.5% eye drops are equivalent to vehicle. Thus healthy volunteers have been selected and have been treated by using a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of either gender, 18 years or older, who were able to give an informed consent
* A score for ocular discomfort of 0-20 mm on the visual analogue scale (VAS) prior to treatment

Exclusion Criteria:

* Known hypersensitivity to any of the constituents of the medications
* Known corticosteroid responder (elevation of intraocular pressure [IOP])
* Known allergic disposition (e.g. hay fever)
* Need of ocular antiallergic treatment
* Wearing of contact lenses
* Any kind of current eye disease (e.g. dry eye)
* Any kind of concomitant ocular treatment
* Any injury or infection in either eye during the last 3 months prior to the first application
* Any medication taken within the last 28 days prior to the first application, except hormonal contraceptives
* Concomitant or previous treatment with antihistamines within a week prior to enrolment
* Pregnant or breast feeding women
* Participation in another clinical study within 4 weeks prior to enrolment
* Hematological diseases such as aplastic anemia, panmyelopathy, or hemolytic icterus; with severe dysfunction of the liver.
* Any medical or laboratory condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the trial per protocol
* Subjects with history of malignancy of any organ system, treated or untreated, within the past five years, whether or not evidence of local recurrence or metastases exist, are excluded, with the exception of localized basal cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-08

PRIMARY OUTCOMES:
Tolerability of the trial drug by evaluating the overall sum-score of the slit lamp examination built by adding up the scores for conjunctival hyperemia, conjunctival edema, palpebral hyperemia, lid edema and corneal edema

SECONDARY OUTCOMES:
Tolerability of the trial drug
and the frequency, severity and relationship to study medication of all adverse events occurring during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis
Locations (1):
- Kopfklinik der Ruprechts-Karls- Universität, Heidelberg, Germany